CLINICAL TRIAL: NCT05964413
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Adaptive Phase III Trial to Investigate Efficacy and Safety of Vilobelimab in the Treatment of Ulcerative Pyoderma Gangrenosum
Brief Title: Phase III Trial to Investigate Efficacy and Safety of Vilobelimab in Ulcerative Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped for futility
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFX-1-P3.4
Record Dates: First submitted 2023-06-29; First posted 2023-07-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — vilobelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vilobelimab (Experimental): Patients will be treated with vilobelimab IV, Q2W for 26 weeks
  Interventions: Drug: vilobelimab
- Placebo (Placebo Comparator): Patients will receive placebo IV in the same schedule as patients in Arm 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vilobelimab — vilobelimab infusion
  Arms: vilobelimab
Drug: Placebo — Placebo Infusion
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, multicenter, adaptive phase III trial to investigate efficacy and safety of vilobelimab in the treatment of ulcerative pyoderma gangrenosum

ELIGIBILITY:
Main Inclusion Criteria:

1. 18 years or older at the time of signing the informed consent.
2. Investigator confirmed clinical diagnosis of ulcerative PG. Diagnosis shall be supported by clinical assessment of PG symptoms via PARACELSUS score (Jockenhofer, Wollina et al. 2019) of 10 points or more (see Appendix - Section 12.1). Note: in case of PARACELSUS score < 10, additional justification shall be provided by the investigator to support clinical diagnosis of ulcerative PG.
3. Minimum of 1 evaluable PG ulcer (other than peristomal) which qualifies as the target ulcer by meeting the following criteria (Orfaly, Reese et al. 2022): area of ≥ 5 cm 2 at screening and baseline

   * circulated by intact skin
   * evaluable by at least 2-dimensional measurement

Main Exclusion Criteria:

1. Patients with target ulcers exceeding 80 cm 2 .
2. Patients with target ulcer in transplanted skin.
3. Surgical wound debridement or negative pressure wound therapy (NPWT) for the target ulcer within 4 weeks before baseline (i.e., start of treatment with IMP).
4. Patient with previous exposure to vilobelimab (IFX-1) prior to baseline (i.e., start of treatment with IMP).
5. Patient receives/has received a vaccine within 2 weeks prior to baseline (i.e., start of treatment with IMP).
6. Any active infection requiring systemic antibiotic or other systemic treatment or suppressive anti-infective therapy within 2 weeks prior to baseline (i.e., start of treatment with IMP).
7. Patients received any systemic medical treatment for PG within 4 weeks prior to baseline
8. Patients received any biological or immunomodulatory therapy for PG within 4 weeks prior to baseline (i.e., start of treatment with IMP), except existing biologic or immunomodulatory therapy used for an underlying disease (other than PG at a stable therapy with no dose adjustments for at least two maintenance doses prior to screening this is allowed to be continued.
9. Patients receiving corticosteroids treatment for PG of more than 10 mg/day of prednisone or equivalent within 4 weeks prior to baseline (i.e., start of treatment with IMP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment with vilobelimab compared to placebo | Week 1 to Week 26
  Efficacy of Vilobelimab compared to placebo - complete closure of the ulcer

SECONDARY OUTCOMES:
Efficacy of treatment with vilobelimab compared to placebo | 2 weeks between study visits
  Proportion of patients achieving disease remission up to and including EOT visit; where disease remission is assessed by the investigator as complete re-epithelization (defined as wound covered by epithelial skin layer or scar) of all PG ulcers, without drainage or dressing requirements
Pain reduction | Week 10 through study completion
  Proportion of patients achieving a pain reduction related to the target ulcer of at least 3 points compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alex GO Loayza, Prof, MD, Principal Investigator — university
Locations (50):
- United States (12):
  - Aby´s New Generation Research, Inc, Hialeah, Florida
  - Dermatology/University of Miami Hospital, Miami, Florida
  - University of Central Florida College of Medicine, Orlando, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Brigham and Women´s Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill Department of Dermatology, Chapel Hill, North Carolina
  - Ohio State University Wexner Medical Cente OSU Dermatology West, Columbus, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
- Australia (4):
  - Premier Specialists, Kogarah, NewSouth Wales
  - The Alfred Hospital, Melbourne, Melbourne, Victoria
  - Veracity Clinical Research Pty Ltd as trustee for the MLS Trust, Brisbane
  - Liverpool Hospital, Sydney
- Belgium (2):
  - Hôpitaux Universitaires de Bruxelles, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
- France (4):
  - CHU Toulouse Hospital Larrey, Toulouse, Occitanie
  - Hospital Edouard Herriot, Lyon
  - CHU de Nantes - Clinique dermatologique, Nantes
  - Saint Louis Hospital, Paris
- Germany (13):
  - Universitätshautklinik Tübingen, Tübingen, Baden Würrtemberg
  - Berge Hautklinik, Erlangen, Bavaria
  - Universitätsklinikum Heidelberg, Heidelberg, Bavaria
  - Klinik und Poliklinik für Dermatologie und Allergologie, München, Bavaria
  - University Hospital Würzburg, Department of Dermatology, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt, Klinik für Dermatologie, Frankfurt am Main, Hesse
  - Catholic Clinic Bochum, Department of Dermatology, Bochum, Nordrhein-Westfalia
  - University of Essen, Germany, Essen, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Department of Dermatology, Venereology and Allergology, Berlin, Germany, Berlin
  - University clinic Duesseldorf Department of Dermatology Heinrich-Heine-University Duesseldorf, Düsseldorf
  - Universitätsklinik für Dermatologie und Venerologie der MLU Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Institut für Versorgungsforschung in der Dermatologie und bei Pflegeberufen (IVDP), Hamburg
  - University Hospital Leipzig AöR, Leipzig
- Hungary (3):
  - Department of Dermatology and Allergology, University of Szeged, Szeged, Csongrad-Csanad
  - Department of Dermatology, University of Debrecen, Debrecen, Hadju-Bihar
  - Department of Dermatology, Venerology and Oncodermatology, University of Pécs, Pécs
- Italy (4):
  - IRCCS Policlinico di Sant'Orsola Alma Mater Studiorum - University of Bologna, Bologna
  - Fondazione IRCCS Ca´ Granda Ospedale Maggiore Policlinico SC Dermatologia, Milan
  - Ospedale Santa Chiara, Pisa
  - AOU Città della salute e della scienza, Turin
- Poland (5):
  - Wojewódzki Specjalistyczny Szpital im. Dr Wł. Biegańskiego w Łodzi; Klinika Dermatologii, Dermatologii Dziecięcej i Onkologicznej Uniwersytetu Medycznego, Lodz
  - Department and Clinics of Dermatology, Venereology and Paediatric Dermatology, Medical University of Lublin,, Lublin
  - Klinika Dermatologii, Chorób Przenoszonych Drogą Płciową i Immunologii Klininczej, Miejski Szpital Zespolony w Olsztynie Clinic of Dermatology,, Olsztyn
  - Państwowy Instytut Medyczny CSK MSWiA, Warsaw
  - City Clinic Przychodnia Lekarsko-Psychologiczna ul. Sliczna 13, Wroclaw, Poland, Wroclaw
- Spain (2):
  - Hospital Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
- University Hospital Basel Department of Dermatology at Universitäre Altersmedizin FELIX PLATTER, Basel, Switzerland